CLINICAL TRIAL: NCT07283731
Title: Phase 2 Trial of Zanzalintinib and Pembrolizumab in Select Subtypes of Advanced/Metastatic Soft-tissue Sarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0952; NCI-2025-09246 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-12-12; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Phase 2; Zanzalintinib; Pembrolizumab; Advanced/Metastatic; Soft-Tissue Sarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Treatment with Zanzalintinib + Pembrolizumab
  Interventions: Drug: Zanzalintinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Zanzalintinib — Given by po
Drug: Pembrolizumab — Given by iv

SUMMARY:
To learn if zanzalintinib and pembrolizumab can help to control select subtypes of advanced/metastatic soft-tissue sarcoma (UPS, MFS, HGPS, and HGUS

DETAILED DESCRIPTION:
Primary Objectives

1. To estimate the progression free survival (PFS), defined as the time from enrollment to time of first event (progressive disease per RECIST v.1.1 criteria or death from any cause) after receiving zanzalintinib and pembrolizumab or date of last contact for participants without an event

Secondary Objectives

1. To estimate the progression free rate (progressive disease per RECIST v.1.1 criteria70 or death from any cause after first drug) at 6 months and 1 year
2. To estimate the overall response rate (ORR) as measured by RECIST v1.1 a
3. To describe the toxicity of zanzalintinib and pembrolizumab, defined by the rate of Grade 3 or higher adverse events by CTCAE v5 criteria

ELIGIBILITY:
Eligibility Criteria

* Participants must have histologically or cytologically confirmed undifferentiated pleomorphic sarcoma (UPS), myxofibrosarcoma (MFS), high grade pleomorphic (HGPS) or undifferentiated sarcoma (HGUS).
* Participant ≥ 18 years of age. Because no dosing or adverse event data are currently available on the use of zanzalintinib in combination with pembrolizumab in participants <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%).
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
* At least 4 weeks since prior chemotherapy.
* At least 2 weeks since radiation therapy for bone metastases, any other radiation therapy within 4 weeks before first dose of study treatment. At least 6 weeks since systemic treatment with radionuclides before first dose of study treatment.
* Participants must have adequate organ and marrow function as defined below within 14 days before first dose of study treatment:

absolute neutrophil count ≥1,500/mcL without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection.

platelets ≥100,000/mcL without transfusion within 2 weeks of screening laboratory sample collection.

hemoglobin ≥ 9 g/dL (≥ 90 g/L) without transfusion within 2 weeks prior to screening laboratory sample collection.

international normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.2 x upper limit of normal (ULN ).

total bilirubin ≤ 1.5 x institutional ULN AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN Alkaline phosphatase (ALP) ≤3 × institutional ULN, . For subjects with documented bone metastasis ALP ≤ 5 x ULN.

creatinine ≤ 1.5 x institutional ULN or calculated creatinine clearance ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft Gault equation.

Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol)

* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for at least 4 weeks. Note: Participants must have stopped corticosteroids or be on physiologic corticosteroid replacement therapy (prednisone ≤ 10 mg daily or equivalent).
* Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first three cycles of therapy.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of zanzalintinib and pembrolizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

  o Postmenopausal (no menses in greater than or equal to 12 consecutive months).

  o History of hysterectomy or bilateral salpingo-oophorectomy.

  o Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).

  o History of bilateral tubal ligation or another surgical sterilization procedure.

  o Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.
* Females must not be pregnant.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Women of childbearing potential must comply for the duration of study participation and through 186 days after the last dose of zanzalintinib and 180 days after the last dose of pembrolizumab, whichever date is later. Men must comply for the duration of study participation and through 96 days after the last dose of zanzalintinib or 96 days of pembrolizumab, whichever date is later.
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
* Consent to MD Anderson companion laboratory protocol 2014-0938 for correlative analyses of biopsies obtained in this trial.

Exclusion Criteria

* Prior treatment with immune checkpoint inhibitors (ICIs)
* Prior treatment with zanzalintinib
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible. Additionally, if participants have received radiation therapy within 4 weeks or systemic therapy with radionucleotides within 6 weeks they are not eligible.
* Participants who are receiving any other investigational agents, as well as cytotoxic or biological systemic anticancer therapy including investigational treatments within 4 weeks of initiating study treatment are excluded.
* Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors) and platelet inhibitors (eg, clopidogrel).

  * Allowed anticoagulants are the following:

    1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
    2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.

Note: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.

* Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

Unstable of deteriorating cardiovascular disorders • Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsade's de pointes).

* Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
* Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study treatment.
* Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before first dose of study treatment.

Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.

Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.

o Prior history of myocarditis.

Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

* Tumors invading the GI-tract from external viscera.
* Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis.
* Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and subject is asymptomatic.
* Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
* Known gastric or esophageal varices.
* Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks.

  * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
  * Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed).
  * Tumors invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. Note: Subjects with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior vena cava) may be eligible following Principal Investigator approval.
  * Other clinically significant disorders that would preclude safe study participation.
* Active infection requiring systemic treatment. Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.
* Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
* Malabsorption syndrome.
* Pharmacologically uncompensated, symptomatic hypothyroidism.
* Moderate to severe hepatic impairment (Child-Pugh B or C).
* Requirement for hemodialysis or peritoneal dialysis.
* History of solid organ or allogeneic stem cell transplant.

  * Participants with brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for at least 3 months.
  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to zanzalintinib or pembrolizumab or other agents used in study.
  * Moderate or strong CYP3A4 inhibitors (see section 5.4).
  * Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load and CD4+ T cell count ≥ 200/µL within 6 months are eligible for this trial.
* Note: To be eligible, participants taking CYP inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose. Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider.

  * Participants with psychiatric illness/social situations that would limit compliance with study requirements.
  * Pregnant women are excluded from this study because zanzalintinib has the potential for teratogenic or abortifacient effects based on its mechanism of action. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with zanzalintinib and pembrolizumab, breastfeeding should be discontinued if the mother is treated with either agent. These potential risks may also apply the other agents used in this study.
  * Major surgery (as defined in Appendix 2) within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (ie nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (eg, simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment.

Note: Fresh tumor biopsies should be performed at least 5 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.

• Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per electrocardiogram (ECG) before first dose of study treatment.

Note: Triplicate ECG evaluations one minute apart will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.

* Inability to swallow tablets or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube.
* Another malignancy that requires active therapy and in the opinion of the Investigator would interfere with monitoring of radiologic assessments of response to Investigational Product, within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy. Incidentally diagnosed prostate cancer is allowed if assessed as stage ≤ T2N0M0 and Gleason score ≤ 6.
* Suspected autoimmune disease, or active or prior documented autoimmune disease within the last 2 years.

Note: Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

* Known positive test for tuberculosis infection if supported by clinical or radiographic evidence of disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Free thyroxine (FT4) outside the laboratory normal reference range. Asymptomatic subjects with FT4 abnormalities can be eligible after Principal Investigator approval.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg daily prednisone equivalent) or any other form of immunosuppressive therapy within 2 weeks prior to first dose of study treatment. Inhaled, intranasal, intraarticular, and topical corticosteroids and mineralocorticoids are allowed. Note: Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Transient short-term use of higher doses of systemic corticosteroids for allergic conditions (eg, contrast allergy) is also allowed.
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment.
* Other conditions, which in the opinion of the Investigator, would compromise the safety of the participant or the participant's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-06-02 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Nakazawa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org